CLINICAL TRIAL: NCT07174739
Title: Efficacy of Quantum Molecular Resonance in Neuropathic Corneal Pain and Corneal Nerve Regeneration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-2421
Record Dates: First submitted 2025-09-14; First posted 2025-09-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Neuropathic Corneal Pain
Keywords: neuropathic corneal pain; eye pain; QMR; Quantum Molecular Resonance; Rexon-Eye
MeSH Terms: conditions — Eye Pain | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quantum Molecular Resonance (QMR) Treatment (Experimental): Participants in this arm will receive Quantum Molecular Resonance (QMR) treatment using the Rexon-Eye device for a total of eight sessions, administered once weekly, with each session lasting 30 minutes. The study consists of nine visits in total: one pre-assessment visit, followed by the eight QMR treatment sessions. The efficacy of QMR treatment will be evaluated through various aspects, including in participants' self-reported symptom relief, clinical ocular surface assessments, and IVCM evidence of corneal nerve regeneration.
  Interventions: Device: Quantum Molecular Resonance (QMR) Treatment

INTERVENTIONS:
Device: Quantum Molecular Resonance (QMR) Treatment — Quantum Molecular Resonance (QMR) treatment will be administered using the Rexon-Eye® device (Resono Ophthalmic, Sandrigo, Italy) according to the protocol recommended by the manufacturer. The device features a contact electrode embedded in a mask worn over the participant's closed eyes, and it delivers stimulation to the epidermis of the closed eyelids, extending up to the lid border with an intensity setting of 4-5 on a scale of 0-10. The treatment is non-invasive and painless.

SUMMARY:
The goal of this study is to evaluate whether Quantum Molecular Resonance (QMR) treatment can effectively reduce eye pain and stimulate corneal nerve regeneration in patients with neuropathic corneal pain (NCP). Participants diagnosed with NCP will attend a total of nine study visits, consisting of one baseline assessment and eight QMR treatment sessions. At each visit, participants will undergo a series of clinical examinations to evaluate changes in the ocular surface, corneal nerves, and tear proteins, and will complete questionnaires regarding their symptoms, eye pain, and quality of life. The investigators will compare these outcomes before and after QMR treatment to determine whether QMR treatment alleviates NCP symptoms and enhances ocular surface and corneal nerve health. The investigators hypothesize that QMR treatment will provide notable pain relief, promote corneal nerve regeneration, and improve overall quality of life for NCP patients.

DETAILED DESCRIPTION:
Neuropathic corneal pain (NCP) is a severe and challenging condition resulting from dysfunctional corneal nerves, with a range of non-specific symptoms. Patients with NCP often experience burning, aching, shooting, or stabbing pain without corresponding clinical signs, and the symptoms are typically unresponsive to conventional dry eye treatments. NCP is associated with various conditions, including dry eye disease, diabetic corneal neuropathy, herpes simplex keratitis, recurrent corneal erosion syndrome, radiation keratopathy, trauma, and ocular surgeries such as cataract or refractive procedures. Psychological conditions like depression and anxiety, and chronic pain states such as fibromyalgia and trigeminal neuralgia, predispose patients to NCP. The effects of NCP can range from mild discomfort impacting daily activities to severe symptoms that significantly impair physical and social well-being. Patients with NCP typically show reductions in morphologic metrics, including corneal nerve fiber length and density, which can be assessed using in vivo confocal microscopy (IVCM). In addition, microneuromas, characterized by irregularly shaped enlargements of terminal nerve endings with poorly defined margins and variable hyper-reflectivity on IVCM, are dynamic indicators of corneal neuropathological recovery.

Treatment of NCP is challenging due to its complex and varied pathophysiology, often requiring multiple approaches. Effective management aims to alleviate pain in the short term and address central sensitization in the long term. Management typically involves anti-inflammatories, nerve-regenerating agents, and mental health support, including artificial tears, topical steroids, autologous serum tears, cryopreserved amniotic membrane, and bandage contact lenses. However, these treatments have drawbacks, and many patients experience persistent pain despite these approaches. This highlights a critical need for novel treatment approaches to address the complexity of NCP more effectively.

Quantum Molecular Resonance (QMR) is an innovative technology that utilizes transpalpebral, non-invasive, high-frequency microcurrent electrical stimulation, promoting the natural regeneration of cells. By applying low-power, high-frequency oscillating electrical currents within the range of 4 to 64 megahertz, QMR leverages the resonance effect to optimize energy delivery to biological tissues. Remarkably, this process achieves significant biological responses without increasing tissue temperature. QMR modulates cellular inflammatory responses by down-regulating pro-inflammatory cytokines while simultaneously upregulating anti-inflammatory ones. The energy package delivered by QMR significantly alters intra- and extracellular ions, changing the transmembrane potential and triggering stem cell replication, and leading to asymmetric regeneration of new stem cells. The Rexon-Eye (Resono Ophthalmic, Sandrigo, Italy) is a QMR-based electrotherapy device developed in 2014. It received Conformité Européene marking in 2016 as a medical device for ocular surface disorders and has patents in Italy and Europe, as well as Health Sciences Authority approval in Singapore. The therapy involves applying specialized mask electrodes to the periorbital area for 20-minute sessions, and it stimulates cellular regeneration and reactivates the lacrimal system, particularly in treating dry eye disease. Previous studies have demonstrated a significant reduction in corneal epithelial damage and an improvement in subjective ocular surface symptoms, as measured by the Ocular Surface Disease Index (OSDI) after treatment compared to placebo, with no reported adverse effects. Furthermore, it has been found that electrical stimulation treatments can effectively reduce ocular pain intensity and improve corneal sensitivity.

The investigators aim to evaluate the efficacy of QMR treatment in alleviating symptoms of NCP and promoting corneal nerve regeneration. The underlying molecular mechanisms by which QMR exerts its effects, including its influence on neuroinflammatory pathways and nerve function, will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 21 years of age.
* Regardless of gender (Male/Female).
* Regardless of race (Chinese/Malay/Indian/Eurasian/Others).
* Diagnosed with neuropathic corneal pain based on the following criteria: presence of neuropathic ocular symptoms (burning, stinging, photophobia, pain, severe dryness), absent or minimal slit-lamp findings to explain the symptoms and corneal nerve abnormalities as detected by IVCM (decreased corneal length and density, presence of neuromas).
* Willing to receive all eye examinations in this study.

Exclusion Criteria:

* Pregnant women.
* Participants carrying active implantable devices (e.g., pacemakers and hearing aids).
* Oncologic patients under treatment; patient who underwent ocular surgery in the last month.
* Participants who had ocular infection within 6 months, or active ocular infection or inflammation; any concomitant ocular diseases that could potentially induce ocular pain, such as uveitis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) to measure eye pain severity | From enrollment to the end of treatment at 8 weeks.
  The VAS is used to assess patients' pain progression and to compare pain severity across different time points. The VAS will be used to measure on a scale of 0 to 10, with higher scores indicating greater pain severity. A score below 4 cm is preferred for effective chronic sensation management.
Ocular Pain Assessment Survey (OPAS) questionnaire to evaluate eye pain features | From enrollment to the end of treatment at 8 weeks.
  The Ocular Pain Assessment Survey (OPAS) is a 27-item questionnaire to evaluate the eye pain from 6 dimensions, including pain intensity for the last 24h, pain intensity for the last 2 weeks, non-eye pain intensity, quality of life, aggravating factors, associated factors and symptom relief. Each question was scored on a scale of 0-10, with higher score representing worse pain.
Extend of corneal nerve impairment assessed by IVCM | From enrollment to the end of treatment at 8 weeks.
  IVCM will be used to capture corneal nerve images before and after surgeries. The extend of corneal nerve damage will be quantified using seven nerve parameters by a specialized image analysis software (ACCMetrics software).

SECONDARY OUTCOMES:
Amount of tear production measured by Schirmer's I test | From enrollment to the end of treatment at 8 weeks.
  Schirmer's I test is a diagnostic method used to measure tear production by placing a standard 5 mm wide Test Strips inside the lower lid margin and assessing the amount of tear absorbed over 5 minutes.
Corneal sensitivity measurements assessed by Cochet-Bonnet esthesiometer | From enrollment to the end of treatment at 8 weeks.
  Corneal sensitivity measurements assess the responsiveness of the cornea to external stimuli using a contact Cochet-Bonnet esthesiometer, which employs a retractable nylon filament marked from 0 to 6 cm. The filament is progressively shortened in 0.5 cm increments until the participant perceives the stimulus. The maximum filament length that successfully triggers a response is recorded in centimeters as a measure of corneal sensitivity.
Level of tear film stability | From enrollment to the end of treatment at 8 weeks.
  Tear Break-up time (TBUT) will be measured by determining the time interval between a complete blink and the first appearance of a dry spot on the corneal surface, indicating tear film stability.
National Eye Institute (NEI) Score | From enrollment to the end of treatment at 8 weeks.
  The cornea will be divided into five regions, each scored ranging from 0 (no fluorescein staining) to 3 (severe fluorescein staining) according to the grading scheme. The total NEI score will range from 0 to 15.
Oxford score | From enrollment to the end of treatment at 8 weeks.
  The staining intensity on the ocular surface will be assessed according to the Oxford score scheme: the staining pattern will be graded on a scale from 0 to 5, indicating the intensity from no staining to severe.
Corneal microneuromas morphology profiles | From enrollment to the end of treatment at 8 weeks.
  IVCM will be used to capture images of corneal microneuromas, which are characterized by irregularly shaped enlargements of terminal nerve endings with poorly defined margins and variable hyper-reflectivity. The images containing corneal microneuromas will be manually identified and the total area and perimeter will be quantified using Image J software.
Ocular Surface Disease Index (OSDI) questionnaire to measure eye symptoms and the impact of quality of life | From enrollment to the end of treatment at 8 weeks.
  The OSDI is a 12-item questionnaire that used to assess the eye symptoms and and their impact on vision-related quality of life. The total OSDI score (ranging between 0 and 100) is used for evaluation, with higher scores representing greater severity of symptoms.
Abundance of tear proteins assessed by quantitative proteomic analysis | From enrollment to the end of treatment at 8 weeks.
  Tear fluid samples will be collected by the strips from Schirmer's I test. Quantitative proteomic analysis technique will be used to measure and compare the abundance of proteins across different samples, providing insights into protein expression, functions, and molecular interactions.
Concentration of tear neuromediators assessed by enzyme-linked immunosorbent assay | From enrollment to the end of treatment at 8 weeks.
  Tear fluid samples will be collected by the strips from Schirmer's I test. The neuromediators concentration in all tear samples will be analyzed using the enzyme-linked immunosorbent assay。

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No